CLINICAL TRIAL: NCT04641351
Title: Injection After Arthroscopic Partial Meniscectomy
Brief Title: Corticosteroid Meniscectomy Randomized Trial
Acronym: CoMeT
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Arthritis Foundation (Other)
Responsible Party: Principal Investigator, Kurt Spindler, MD, Grant PI, Arthritis Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-1074
Record Dates: First submitted 2020-10-15; First posted 2020-11-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis, Knee; Meniscus Tear; Meniscus; Degeneration; Synovitis
Keywords: knee pain; arthroscopic partial meniscectomy; post-traumatic OA; patient reported outcome
MeSH Terms: conditions — Osteoarthritis, Knee; Synovitis | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- corticosteroid (Experimental): Triamcinolone extended release (32 mg) administered as an intraarticular injection at the conclusion of arthroscopic partial meniscectomy.
  * Knee injury and Osteoarthritis Outcome Score (KOOS) pain at 6 and 12 months
  * T1ρ and T2 imaging of cartilage and meniscus at 3 and 12 months
  * Morphologic grading of cartilage using the MOAKS score at 3 and 12 months
  * 3D bone shape from MRI Osteoarthritis Knee Score (MOAKS) using statistical shape modeling at 3 and 12 months
  * Improvement in blood, serum and urine inflammatory biomarker profiles at 3 and 12 months
  Interventions: Drug: Zilretta Injectable Product or Placebo
- Placebo (Placebo Comparator): Normal saline of 5 mL administered as an intraarticular injection at the conclusion of arthroscopic partial meniscectomy.
  * KOOS pain at 6 and 12 months
  * T1ρ and T2 imaging of cartilage and meniscus at 3 and 12 months
  * Morphologic grading of cartilage using the MOAKS score at 3 and 12 months
  * 3D bone shape from MRI using statistical shape modeling at 3 and 12 months
  * Improvement in blood, serum and urine inflammatory biomarker profiles at 3 and 12 months
  Interventions: Drug: Zilretta Injectable Product or Placebo

INTERVENTIONS:
Drug: Zilretta Injectable Product or Placebo — The purpose of this intervention is to determine the use of extended release steroid knee injection (Zilretta) at the end of the surgery and its effects on your knee pain.In this study Zilretta will be injected intra-operatively for your arthroscopic partial meniscectomy (APM) surgery.Participants will have MRIs x-rays, and provide a sample of the synovial fluid from both knees at the beginning of surgery. This fluid is drained at the beginning of surgery and then usually discarded. Three samples each of blood and urine will be collected over the study period from each participant and sample of joint (synovial tissue) taken. Participants will be asked to answer questions about knee pain.
  Other Names: triamcinolone acetonide

SUMMARY:
Synovitis has an important role in the symptoms and progression of Osteoarthritis (OA). Inflamed synovium has been associated with both increased symptoms and increased progression in OA patients. Furthermore, synovitis observed during knee arthroscopy in our patients undergoing arthroscopic partial meniscectomy (APM) was associated with worse symptoms while adjusting for confounding factors.Therefore, a better understanding of synovitis as a predictor of outcome after APM and as a target for treatment is needed to improve outcomes in this patient population.

Triamcinolone has been shown to decrease synovitis-associated outcomes in both animal and human studies after anterior cruciate ligament (ACL) injury. In a porcine model of ACL injury, treatment with triamcinolone resulted in decreased formation of synovitis-related collagen breakdown products as well as decreased cellularity of the synovium.And in a trial of triamcinolone injected after ACL injury, similar findings of decreased C-telopeptide of type II collagen (CTX-II), associated with collagen type II breakdown, was found in knees administered triamcinolone compared to placebo controls.

DETAILED DESCRIPTION:
Symptomatic meniscal tear with pain and mechanical symptoms of catching and locking ,a phenotype of early OA, and often prompts patients who have failed physical therapy to elect APM to improve their symptoms. This arthroscopic surgery presents a unique opportunity to evaluate the intraarticular status of the joint including joint fluid biomarkers and synovial tissue for signs of inflammation in patients with mild to moderate OA. Since no post-op tissue repair is desired after APM, in contrast to other post-traumatic OA (PTOA) models such as anterior cruciate ligament reconstruction, the APM cohort can be used to test novel interventions to slow down PTOA development by suppressing synovitis and inflammation. Results from this trial in this patient population could be applied to the broader population of many millions of patients with mild to moderate OA who never undergo arthroscopy.

There are currently approximately 1,000,000 APMs performed in the United States each year, and about 70 percent of patients have a clinically significant improvement in symptoms after surgery. Much of this variation in outcome is unexplained but is hypothesized to be related to synovitis and joint inflammation that is currently unmeasured and untreated in usual clinical care.

This is a randomized controlled trial of extended release triamcinolone for efficacy to improve patient reported outcome measures after APM. The investigators will evaluate joint fluid and synovial tissue biomarkers to assess joint inflammation as a predictor of treatment response, use quantitative 3T MRI to evaluate cartilage and meniscus composition and 3D bone shape, which are sensitive imaging markers for early joint degeneration, and use a prospective surgical episode data collection system to capture patient reported outcomes and surgeon reported operative data.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 40 and older
2. Scheduled for APM with enrolling surgeon
3. Arthroscopic evidence of structural OA including at least one surface with grade 2 chondral change
4. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Females who are pregnant or nursing or plan to become pregnant during the study; men who plan to inseminate a partner or donate sperm
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
3. Known or suspected hypersensitivity to Zilretta (or component of Zilretta) or triamcinolone acetonide
4. Kellgren and Lawrence Grade IV (severe OA; arthroplasty is typically preferred over APM in this setting)
5. Injection with corticosteroid into affected knee in past 12 weeks
6. Injection with platelet rich plasma into affected knee in past 12 weeks
7. Injection with hyaluronic acid into affected knee in past 24 weeks
8. Plan for cartilage resurfacing procedure (microfracture, autologous chondrocyte implantation, osteochondral autograft or allograft), ligament reconstruction or other open procedure
9. Bilateral surgery
10. Unable to undergo MRI due to implanted medical device, aneurysm clamp, metal fragments in eye, etc.
11. Absence of at least one area of grade 2 chondral change on diagnostic arthroscopy (patients without structural OA are excluded)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Knee injury and Osteoarthritis Outcome Score (KOOS) from baseline and 3 months. | 0 and 3 months
  Knee pain of participants; a higher score represents a desired outcome; zero representing extreme knee problems and 100 representing no knee problems

SECONDARY OUTCOMES:
Change in Knee injury and Osteoarthritis Outcome Score (KOOS) from baseline, 6 and 12 months. | 0, 6, and 12 months
  Knee pain of participants; a higher score represents a desired outcome; zero representing extreme knee problems and 100 representing no knee problems
Change in Inflammatory biomarkers in circulation from baseline, 3 and 12 months. | 0, 3, and 12 months
  Urine; CTX-II
Change in Inflammatory biomarkers of the knee joint from baseline, 3, and 12 months. | 0, 3, and 12 months
  The increase or decrease from the combination of following markers in the Synovial fluid will help characterize the profile of knee joint; TGF-ß1, neutrophil elastase, IL-1, IL-6, IL-8, TNF, MCP-1, MIP1, MMP-3, MMP-10, MMP activity, sGAG, aggrecanase, TIMP-1, and PGE2
Change in Inflammatory biomarkers in circulation from baseline, 3 and 12 months. | 0, 3 and 12 months
  The increase or decrease from the combination of the following markers in the serum will help characterize the inflammatory profile of the individual systemically; hyaluronic acid, IL-1, IL-6, IL-8, TNF, TIMP-1, MMP-10, MCP-1, MIP1, and PGE2
Change in Magnetic Resonance Imaging relaxation time (milliseconds of T1 and T2) from baseline, 3, and 12 months. | 0, 3 and 12 months
  Quantitative measurement of cartilage, longer relaxation time represents a poor outcome
Change in Whole-Organ Magnetic Resonance Imaging Score (WORMS) from baseline, 3, and 12 months. | 0, 3 and 12 months
  Bone shape, a higher score represents a poor outcome; zero representing no knee problems and 332 representing knee problems
Change in Magnetic Resonance Imaging morphological grading from baseline, 3, and 12 months. | 0, 3 and 12 months
  Modified MRI Osteoarthritis Knee Score (MOAKS); a higher score represents a poor outcome; zero representing no knee problems and 332 representing knee problems

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Jones, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Bringham and Women's Hospital, Boston, Massachusetts
  - Cleveland Clinic Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No